CLINICAL TRIAL: NCT01633775
Title: Re-Trabeculectomy Versus Ahmed Glaucoma Valve Implantation in Secondary Surgical Management of Patients With Refractory Primary Open Angle Glaucoma: a Three-year Comparative Study
Brief Title: Re-Trabeculectomy Versus Ahmed Glaucoma Valve Implantation in Secondary Surgical Management of Patients With Refractory Glaucoma
Status: Completed | Type: Observational
Sponsor: Vanak Eye Surgery Center (Other)
Responsible Party: Principal Investigator, Nariman Nassiri, Prinicpal Investigator, Vanak Eye Surgery Center
Other Study IDs: VESC#2007-056
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-06

CONDITIONS: Refractory Primary Open Angle Glaucoma
Keywords: Refractory primary open angle glaucoma; trabeculectomy; ahmed valve implant
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ahmed glaucoma implant
  Interventions: Procedure: Implantation of Ahmed glaucoma tube shunt, and Trabeculectomy with MMC
- Trabeculectomy with mitomycin C (MMC)
  Interventions: Procedure: Implantation of Ahmed glaucoma tube shunt, and Trabeculectomy with MMC

INTERVENTIONS:
Procedure: Implantation of Ahmed glaucoma tube shunt, and Trabeculectomy with MMC — In the Ahmed implant group, the tube shunts used were the valved 184-mm2 surface area (Model FP7; New World Medical, Inc, Rancho Cucamonga, California, USA). In the Trabeculectomy group, a routine trabeculectomy surgery was performed.

SUMMARY:
The purpose of this study is to compare three-year outcomes of re-trabeculectomy with those of Ahmed glaucoma valve implantation in secondary surgical management of patients with primary open angle glaucoma (POAG) and a history of previous failed trabeculectomy.

DETAILED DESCRIPTION:
Currently, lowering intraocular pressure (IOP) is the only treatment modality to prevent or slow progression of glaucomatous optic nerve damage. Incisional procedures are indicated when medical therapy and/or laser procedures cannot adequately reduce IOP. Trabeculectomy is the most common glaucoma incisional procedure globally. On the other hand, glaucoma drainage devices that have been historically reserved for cases of glaucoma deemed at high risk of failure have increasingly gained popularity particularly in eyes with previous history of glaucoma surgery.

There is still no agreement on the appropriate surgical procedure in those with prior glaucoma surgery. The five-year tube versus trabeculectomy (TVT) study, which evaluated the efficacy and safety of Baerveldt glaucoma implant versus trabeculectomy, showed that both surgical procedures had similar IOP reduction and use of anti-glaucoma medication; tube shunt surgery had a higher success rate than trabeculectomy with mitomycin C (MMC); the trabeculectomy/MMC had higher incidence of early postoperative complications compared to tube shunt surgery; and rates of late postoperative complications, reoperation for complications, and cataract extraction were comparable in both treatment groups.

In this study, the investigators compared three-year outcomes of re-trabeculectomy with those of Ahmed glaucoma valve implantation in secondary surgical management of patients with primary open angle glaucoma and a previous history of failed trabeculectomy.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled glaucoma defined as (1) IOP not achieving previously assigned target pressure despite prior trabeculectomy and use of maximally tolerated anti-glaucoma medication; and (2) recent progression of the disease based on glaucomatous changes in optic disc appearance and/or worsening of the visual field exam.
* In the case of two eligible eyes, only the first eye being operated on was enrolled

Exclusion Criteria:

* Younger than 40 years old
* Visual acuity of no light perception
* Lens opacity
* Elevated IOP associated with silicone oil
* Prior ocular surgeries other than one trabeculectomy with MMC
* Previous cyclodestructive treatment
* Increased risk of endophthalmitis
* Posterior segment disorders
* Pre-existing ocular comorbidities (e.g. pterygium,phacodonesis,corneal opacity, or corneal endothelial dystrophies)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory primary open angle glaucoma and a history of failed trabeculectomy with mitomycin C (MMC).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in target intraocular pressure (IOP) | day 1, week 1, months 1,3,6,9,12,18,24,30,36
  All patients had a target IOP that had been assigned for them by the same surgeon prior to their initial failed trabeculectomy/MMC. The routine practice of the surgeon has been to set target IOP based on the Best Practice Treatment Algorithm for POAG. This was based on at least 25% reduction in baseline IOP. Target IOP needs constant reevaluation during the follow-up based on disease progression. In our study, success and failure were considered to be assessed based on change in the target pressure.

SECONDARY OUTCOMES:
Number of anit-glaucoma medications | day 1, week 1, months 1,3,6,9,12,18,24,30,36
Visual Acuity | day 1, week 1, months 1,3,6,9,12,18,24,30,36
Mean deviation of visual field exam | Months 6,12,18,24,30,36
  Only visual field results where consecutive field tests did not show an improvement of 2 dB or more in the mean deviation (MD) over the baseline reading were included as we considered the phenomenon of learning effect in our analysis.
Surgical Success | day 1, week 1, months 1,3,6,9,12,18,24,30,36
  Surgical failure was defined as persistent IOP of more than target pressure on maximally tolerated medications or IOP less than 6 mm Hg on two consecutive visits, phthisis bulbi, reduction of vision to no light perception, removal of the shunt implant, reoperation for glaucoma, or any devastating intraoperative and postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Nariman Nassiri, MD, MPH, Principal Investigator — Vanak Eye Surgery Center
Locations (3):
- Iran (3):
  - Imam Hossein Medical Center, Tehran
  - Negah Eye Hospital, Tehran
  - Vanak Eye Surgery Center, Tehran

REFERENCES:
- [Background] Ramulu PY, Corcoran KJ, Corcoran SL, Robin AL. Utilization of various glaucoma surgeries and procedures in Medicare beneficiaries from 1995 to 2004. Ophthalmology. 2007 Dec;114(12):2265-70. doi: 10.1016/j.ophtha.2007.02.005. Epub 2007 Apr 27. PMID 17466376
- [Background] Chen PP, Yamamoto T, Sawada A, Parrish RK 2nd, Kitazawa Y. Use of antifibrosis agents and glaucoma drainage devices in the American and Japanese Glaucoma Societies. J Glaucoma. 1997 Jun;6(3):192-6. PMID 9211144
- [Background] Joshi AB, Parrish RK 2nd, Feuer WF. 2002 survey of the American Glaucoma Society: practice preferences for glaucoma surgery and antifibrotic use. J Glaucoma. 2005 Apr;14(2):172-4. doi: 10.1097/01.ijg.0000151684.12033.4d. PMID 15741822
- [Background] Gedde SJ, Schiffman JC, Feuer WJ, Parrish RK 2nd, Heuer DK, Brandt JD; Tube Versus Trabeculectomy Study Group. The tube versus trabeculectomy study: design and baseline characteristics of study patients. Am J Ophthalmol. 2005 Aug;140(2):275-87. doi: 10.1016/j.ajo.2005.03.031. PMID 16086949
- [Background] Gedde SJ, Schiffman JC, Feuer WJ, Herndon LW, Brandt JD, Budenz DL. Treatment outcomes in the tube versus trabeculectomy study after one year of follow-up. Am J Ophthalmol. 2007 Jan;143(1):9-22. doi: 10.1016/j.ajo.2006.07.020. Epub 2006 Sep 1. PMID 17083910
- [Background] Gedde SJ, Herndon LW, Brandt JD, Budenz DL, Feuer WJ, Schiffman JC. Surgical complications in the Tube Versus Trabeculectomy Study during the first year of follow-up. Am J Ophthalmol. 2007 Jan;143(1):23-31. doi: 10.1016/j.ajo.2006.07.022. Epub 2006 Sep 1. PMID 17054896
- [Background] Gedde SJ, Schiffman JC, Feuer WJ, Herndon LW, Brandt JD, Budenz DL; Tube Versus Trabeculectomy Study Group. Three-year follow-up of the tube versus trabeculectomy study. Am J Ophthalmol. 2009 Nov;148(5):670-84. doi: 10.1016/j.ajo.2009.06.018. Epub 2009 Aug 11. PMID 19674729
- [Background] Gedde SJ, Schiffman JC, Feuer WJ, Herndon LW, Brandt JD, Budenz DL; Tube versus Trabeculectomy Study Group. Treatment outcomes in the Tube Versus Trabeculectomy (TVT) study after five years of follow-up. Am J Ophthalmol. 2012 May;153(5):789-803.e2. doi: 10.1016/j.ajo.2011.10.026. Epub 2012 Jan 15. PMID 22245458
- [Background] Gedde SJ, Herndon LW, Brandt JD, Budenz DL, Feuer WJ, Schiffman JC; Tube Versus Trabeculectomy Study Group. Postoperative complications in the Tube Versus Trabeculectomy (TVT) study during five years of follow-up. Am J Ophthalmol. 2012 May;153(5):804-814.e1. doi: 10.1016/j.ajo.2011.10.024. Epub 2012 Jan 14. PMID 22244522
- [Background] Serle J, Cantor L, Gross R, Katz J, Mundorf T, Noecker R, Severin T, Simmons S, Walt J, Casciano J, Evans S, Doyle J. Best practice treatment algorithm for primary open-angle glaucoma: implications for U.S. ophthalmology practice. Manag Care Interface. 2002 Jul;15(7):37-48. PMID 12143296
- [Background] Huang MC, Netland PA, Coleman AL, Siegner SW, Moster MR, Hill RA. Intermediate-term clinical experience with the Ahmed Glaucoma Valve implant. Am J Ophthalmol. 1999 Jan;127(1):27-33. doi: 10.1016/s0002-9394(98)00394-8. PMID 9932995
- [Background] Wilson MR, Mendis U, Smith SD, Paliwal A. Ahmed glaucoma valve implant vs trabeculectomy in the surgical treatment of glaucoma: a randomized clinical trial. Am J Ophthalmol. 2000 Sep;130(3):267-73. doi: 10.1016/s0002-9394(00)00473-6. PMID 11020403
- [Background] Topouzis F, Coleman AL, Choplin N, Bethlem MM, Hill R, Yu F, Panek WC, Wilson MR. Follow-up of the original cohort with the Ahmed glaucoma valve implant. Am J Ophthalmol. 1999 Aug;128(2):198-204. doi: 10.1016/s0002-9394(99)00080-x. PMID 10458176
- [Background] Wilson MR, Mendis U, Paliwal A, Haynatzka V. Long-term follow-up of primary glaucoma surgery with Ahmed glaucoma valve implant versus trabeculectomy. Am J Ophthalmol. 2003 Sep;136(3):464-70. doi: 10.1016/s0002-9394(03)00239-3. PMID 12967799
- See also: Primary Open Angle Glaucoma Preferred Practice Pattern — http://one.aao.org/CE/PracticeGuidelines/PPP.aspx?sid=ca9ec1b5-2567-4e85-96f6-b6540e5ac5a1